CLINICAL TRIAL: NCT03258320
Title: A Phase II-III Study of Neoadjuvant Chemotherapy Involving Cabazitaxel, Docetaxel, Mitoxantrone or Satraplatin (CDMS) Followed by Surgery for Patients With High Risk Prostate Cancer
Brief Title: A Randomised Trial of Cabazitaxel, Docetaxel, Mitoxantrone or Satraplatin (CDMS) Plus Surgery for Prostate Cancer Patients
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Fudan University (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Yu Sun, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCA-81472709
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer Patients
Keywords: Cabazitaxel; Docetaxel; Mitoxantrone; Satraplatin; Surgery; Prostate Cancer; Localized; High Risk
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; Docetaxel; Mitoxantrone; satraplatin

STUDY DESIGN:
Intervention Model Description: Chemotherapy (single agent of CDMS) will be performed 45 days before surgery for patients who are diagnosed with prostate cancer without severe distant metastasis. The chemotherapy using CDMS will be done for 4 cycles within 30 days after first diagnosis of prostate cancer.
Who Masked: Participant, Care Provider
Masking Description: Both the participants and care providers will be blind to the agents, but the investigators will be aware of and keep track of the whole regime and agents.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDMS, Surgery (Experimental): Preoperative chemotherapy using Cabazitaxel, Docetaxel, Mitoxantrone or Satraplatin (CDMS) as a single agent performed 45 days before surgery：Cabazitaxel 25 mg/m2, Docetaxel 35 mg/m2, Mitoxantrone 4 mg/m2 or Satraplatin 80 mg/m2, through intravenous (IV) or oral (Satraplatin) administration. IV or oral administration once every 7 days, totally 4 cycles. There is a 17-day interval between the last dose and surgery.
  Procedure: radical prostatectomy surgery.
  Interventions: Drug: Cabazitaxel, Docetaxel, Mitoxantrone or Satraplatin
- Control (No Intervention): No neoadjuvant chemotherapy using CDMS will be done for patients who are diagnosed with localized prostate cancer but subject to direct surgery to radically remove the primary tumor.

INTERVENTIONS:
Drug: Cabazitaxel, Docetaxel, Mitoxantrone or Satraplatin — As preoperative neoadjuvant chemotherapy, drugss including Cabazitaxel, Docetaxel, Mitoxantrone or Satraplatin (CDMS) will be administered as a single agent performed 45 days before surgery：Cabazitaxel 25 mg/m2, Docetaxel 35 mg/m2, Mitoxantrone 4 mg/m2 or Satraplatin 80 mg/m2, through intravenous (IV) or oral (Satraplatin) administration. IV or oral administration once every 7 days, totally 4 cycles. There is a 17-day interval between the last dose and surgery.
  Other Names: Jevtana, Taxotere, Novantrone, JM216.
  Arms: CDMS, Surgery

SUMMARY:
Current agents administered in therapeutic regimens of prostate cancer employ different mechanisms to eliminate neoplastic cells by inducing substantial apoptosis and causing tumor regression. Treatment with neoadjuvant chemotherapy before radical prostatectomy may better control the tumor before it has the chance to convert into the disease of castration-resistant prostate cancer (CRPC), which is finally refractory to most modalities of clinical intervention with a clinically lethal nature.

DETAILED DESCRIPTION:
Prostate cancer is the development of neoplasia in the prostate, a major gland in the male reproductive system. While most prostate cancers grow slowly, some can develop relatively quickly and aggressively. In a later stage of the disease, cancer cells may disseminate from the prostate to other organs of the body, particularly the bone, lung, brain and lymph node. Prostate cancer initially cause no symptoms, but in an advanced stage it can cause difficulty in urinating, blood in the urine, or pain in the pelvis. A non-malignant or precursor form of prostate cancer known as benign prostatic hyperplasia may produce similar symptoms, although it is essentially not invasive.

Many prostate cancer patients can be safely followed with active surveillance or watchful actions. However, the major forms of clinical treatments include a combination of surgery, radiation, hormone therapy or chemotherapy. If it only occurs inside the prostate, the disease is generally curable. However, when cancer cells have spread to the bones, cytotoxic or harsh therapies are necessary. Outcomes depend on a person's age and other health conditions as well as how aggressive and extensive the cancer is. Most people with prostate cancer do not end up dying from the disease, and the 5-year survival rate in the United States is approximately 99%. To date, it is the 2nd most common type of malignancy and the 5th leading cause of cancer-related death in men. In 2012 it affected 1.1 million men and claimed 307,000 deaths. Prostate cancer occur more frequently in the western countries or developed world, but incidence rates have been continuously arising in the developing countries. Clinical detection increased significantly in the 1980s and 1990s in the global range due to development of the gold standard--PSA testing. Studies of males who died from unrelated causes have found prostate cancer in 30% to 70% of those over the age of 60.

Most hormone-naive prostate cancers become resistant to treatments after 1-3 years and resume growth despite hormone therapy, a condition termed as "hormone-refractory prostate cancer" (HRPC) or "castration-resistant prostate cancer (CRPC)". The most prevalent chemotherapeutic agent docetaxel (Taxotere) has been used as a standardized modality for CRPC and provides a median survival benefit of 2-3 months. A second-line chemotherapy involves cabazitaxel. Although combination of bevacizumab, docetaxel, thalidomide and prednisone appears effective in the treatment of CRPC, these agents are usually used after the occurrence of CRPC, not before. Thus, whether or not these patients should receive chemotherapy prior to development of CRPC, and whether this approach can prevent the aggressive progression of the disease to a treatment refractory status, remain largely open but intriguing questions.

In this study, investigators performed a Phase I, single agent exploration, multicenter clinical trial to establish the treatment efficacy of several chemotherapeutic agents in patients with high risk localized prostate cancer who have developed the primary cancer in prostate. Up to 5 cohorts have been enrolled to determine the effectiveness and safety of single therapeutic strategy. Besides the five-year disease-free survival, overall survival and five-year metastasis-free survival post treatment, investigators also take into account the anticancer agent-induced tumor stroma damage extent, which may provide further evidence to support the treatment efficacy and assess the potential influence of a damaged tumor microenvironment on disease progression or regression in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* 40 ≤ age ≤ 75 years with histologically proven PCa
* no severe major organ dysfunction
* WHO performance status of 0 or 1
* no prior cancer chemotherapy
* A Clinical Stage ≥ T2c (T2c, N0, M0) of prostate cancer but ideally without diagnosed distant metastasis (according to the 2016 American Joint Committee on Cancer (AJCC) definition of TNM staging system, Staging Manual, Eighth Edition) as determined by a preoperative evaluation that included a pleural computed tomography (CT) scan.

Exclusion Criteria:

* age ≥ 76
* severe major organ dysfunction
* WHO performance status of >1
* prior cancer chemotherapy
* Stage IV.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All participant patients should be male, adult.
Enrollment: 300 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
5 years disease-free survival | 5 years
  There is no disease-associated progression during the 5 years post treatment (chemotherapy plus surgery).

SECONDARY OUTCOMES:
5 years overall survival and metastasis-free survival | 5 years
  The overall survival status and distant metastasis-free survival status during the 5 years post treatment (chemotherapy plus surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Yu Sun, Ph.D, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Qilu Hospital of Shandong University, Qingdao, Shandong
  - Zhongshan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No
Investigators are happy to make individual participant data (IPD) available to other researchers upon request, as long as the data are not confidential and not restrained by the ethics policy.